CLINICAL TRIAL: NCT04076475
Title: Effects of Neuromuscular Electrical Stimulation on Patients With Prolonged Mechanical Ventilation
Brief Title: Neuromuscular Electrical Stimulation in Patients With Prolonged Mechanical Ventilation
Acronym: NMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chen Yen-Huey, assist professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201802160A3
Record Dates: First submitted 2019-08-29; First posted 2019-09-03 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-02

CONDITIONS: Prolonged Mechanical Ventilation
Keywords: neuromuscular electrical stimulation; tissue oxygenation; prolonged mechanical ventilation; metabolic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electrical stimulation (Experimental): receive daily NMES for 30 min/session for 10 days.
  Interventions: Device: neuromuscular electrical stimulation
- Control (Sham Comparator): receive similar electrical stimulation (ES) procedure as those in the intervention group but with ES machine power off.
  Interventions: Device: neuromuscular electrical stimulation

INTERVENTIONS:
Device: neuromuscular electrical stimulation — Participants will receive muscular electrical stimulation on quadriceps muscle and abdominal muscles for 30 min/day for 10 days

SUMMARY:
Prolonged mechanical ventilation has been defined as the need for >21 days. The muscle weakness occurred most commonly in patients with PMV and resulted in increasing time to wean from mechanical ventilation, and longer stay in hospital.

Neuromuscular electrical stimulation (NMES) involves applying a stimuli to skeletal muscle, to trigger muscle contraction, and it can be used for the recovery of muscle mass and muscle strength following prolonged immobilization. NMES also improve microcirculation and systemic circulation in patients with cardiopulmonary diseases.

The purposes of this study:

1. to examine the acute effects of NMES on the microcirculation, physiologic response and metabolic demand in patients with PMV.
2. to investigate the training effects of NMES on microcirculation, muscle strength and weaning outcomes in patients with PMV.

METHODS: Subjects with PMV are recruited and are randomly assigned into NMES (n=20) or control group (n=20).The NMES group receive daily NMES for 30 min/session for 10 days. The assessment of muscle strength and weaning profile were performed before and after intervention. During the first and the last NMES session, the status of microcirculation and local muscle tissue oxygenation will be measured by NIRS, and the metabolic status will be measured by IC. The ventilator weaning rate and length of stay in RCC will be recorded.

DETAILED DESCRIPTION:
Scientific and technologic advances in medicine have resulted in the ability of the medical team to prolong life. One consequence of life-extending advancements in technology is the increasing numbers of patients requiring prolonged mechanical ventilation (PMV). Prolonged mechanical ventilation has been defined as the need for 21 days, of consecutive mechanical ventilation for six hours/day. The interaction of underlying diseases and prolong bedridden result in various complication in patients with PMV. Known complications can include: muscle weakness, atelectasis, and deconditioning. The muscle weakness occurred most commonly in patients with PMV and resulted in increasing time to wean successfully from mechanical ventilation, and longer stay in hospital. Exercise is effective in improving muscle strength and physical function in patients with heart failure and chronic obstructive pulmonary disease (COPD. However, patients with PMV may be too fragile to perform excise. Neuromuscular electrical stimulation (NMES) involves applying a series of stimuli to skeletal muscle, primarily to trigger muscle contraction, and it can be used for the recovery of muscle mass and muscle strength following prolonged immobilization. NMES also improve microcirculation and systemic circulation in patients with cardiopulmonary diseases. In addition, the application of NMES increases oxygen consumption of whole body and elicits physiologic effects that are similar to aerobic exercise. However, the effects of NMES on the PMV population remain unclear. Near-infrared spectroscopy (NIRS) is a recently developed noninvasive method of measuring tissue oxygenation, blood flow, and local tissue metabolism. NIRS combined with a vascular occlusion test is proposed as a tool to assess the microvascular response. Indirect calorimetry (IC) uses the method of breath-bybreath monitoring by pneumotachography to measure oxygen consumption (VO2) and carbon dioxide production (VCO2).

The purposes of this study:

1. to examine the acute effects of NMES on the microcirculation, physiologic response and metabolic demand in patients with PMV.
2. to investigate the training effects of NMES on microcirculation, muscle strength and weaning outcomes in patients with PMV. METHODS: Subjects who have been on ventilator for>= 21 days are recruited form respiratory care center (RCC) and are randomly assigned into NMES (n=20) or control group (n=20).The NMES group receive daily NMES for 30 min/session for 10 days. The assessment of muscle strength and weaning profile were performed before and after intervention. During the first and the last NMES session, the status of microcirculation and local muscle tissue oxygenation will be measured by NIRS, and the metabolic status will be measured by IC. The mechanical ventilator weaning outcomes and length of stay in RCC will be recorded. The results of this study help us to confirm whether the application of NMES is beneficial in the improvement of muscle strength in patients with PMV, and to furtherly understand the mechanisms. The results may provide an alternative options for clinicians functional and hospitalization outcomes in patients with PMV.

ELIGIBILITY:
Inclusion Criteria:

1. age ≧ 20 years;
2. MV for > 6 h/day for > 21 days; and
3. medical stability, absence of signs and symptoms of infection, and hemodynamic stability).
4. hemodynamic stable without or with a low dose of vasopressor ((Dopamine or Dobutamine <5μg/kg/min)

Exclusion Criteria:

1. acute lung or systemic infection,
2. ongoing neuromuscular disease (e.g., myasthenia gravis, Guillain-Barre disease)
3. bone contracture or skin lesion
4. obesity [body mass index (BMI) >35 kg/m2].
5. disease at end-stage with expecting survival <=6month
6. pregnancy
7. severe edema (deep indentation when pressing a finger into the skin, requiring >30 s to rebound

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
tissue oxygenation | the 1st day of intervention
  local muscle tissue oxygenation
tissue oxygenation | the 10th day of intervention
  local muscle tissue oxygenation
muscle strength | the 1st day of intervention
  Medical research council score. The score ranges from a 0 points (zero strength) to 5 points (good)
muscle strength | the 10th day of intervention
  Medical research council score. The score ranges from a 0 points (zero strength) to 5 points (good).
pulmonary function (maximal inspiratory pressure) | the 1st day of intervention
  pressure gauge
pulmonary function (maximal inspiratory pressure) | the 10th day of intervention
  pressure gauge
oxygen consumption | the 1st day of intervention
  the amount of oxygen that body consume, is measured by indirect calorimetry
oxygen consumption | the 10th day of intervention
  the amount of oxygen that body consume, is measured by indirect calorimetry
energy expenditure (calories) | the 1st day of intervention
  the amount of energy expenditure which is measured by indirect calorimetry
energy expenditure (calories) | the 10th day of intervention
  the amount of energy expenditure which is measured by indirect calorimetry
pulmonary function (rapid shallow breathing index) | the 1st day of intervention
  respiratory rate/tidal volume
pulmonary function (rapid shallow breathing index) | the 10th day of intervention
  respiratory rate/tidal volume

SECONDARY OUTCOMES:
weaning rate | through study completion, an maximal 42 days
  ventilator weaning results (weaning successful/failure)
length of stay in respiratory care center | through study completion, an maximal 42 days
  the total days of stay in respiratory care center

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Huey Chen, PhD, Principal Investigator — Chang Gung University
Locations (2):
- Taiwan (2):
  - Chang Gung University, Taoyuan
  - Dept of Respiratory therapy, Chang Gung University, Taoyuan District

IPD SHARING:
Plan to Share IPD: No